CLINICAL TRIAL: NCT03951727
Title: Long Superficial Femoral Artery Stenting With SuperA Interwoven Nitinol Stents - Siberia
Brief Title: Stella Supera Siberia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSK001
Record Dates: First submitted 2019-04-24; First posted 2019-05-15 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Atherosclerosis; Peripheral Arterial Disease; Superficial Femoral Artery Occlusion
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular treatment for PAD (Other): Single group study (1 arm)
  Interventions: Device: Endovascular treatment for PAD

INTERVENTIONS:
Device: Endovascular treatment for PAD — Long femoropopliteal stenting with SuperA devices

SUMMARY:
Endovascular treatment with stenting is currently used in the treatment of femoro-popliteal lesions. This technique tends to extend to lesions for which the gold standard remains until now the open surgery treatment (lesions TASC C and D).

The primary objective of the study was to evaluate the clinical efficacy at 12 months of the SuperA stent (Abbott) in the treatment of long de novo atherosclerotic lesions TASC C and D in patients with symptomatic peripheral arterial disease. The secondary objectives are to evaluate the clinical effectiveness of the SuperA stent at 24 months, according to clinical, morphological and haemodynamic criterias, the possible influence of calcifications and the quality of life of patients

DETAILED DESCRIPTION:
Patient will be recruiting during 1 year. Patient will be followed in the study during 2 years. Pre-operative exams are collected. Patients are asked to give their oral authorization to participate in the study by their surgeon.

Patient can be included up to the next day of the intervention.

Endovascular treatment of femoropopliteal lesion with SuperA stents :

Intervention will be achieved in operative room, under local anesthesia and sedation or general anesthesia. An angio-CT or an arteriography is necessary to attest the presence for TASC C or D lesion involving the superficial femoral and/or popliteal arteries.

The long femoropopliteal lesion must be pre-dilated during 3 minutes with a balloon of 1mm diameter more than the stent to be implanted.

A control arteriography will be done before the implantation of the stent and at the end of the intervention to assess the success of the procedure.

If needed, endovascular treatment could be realized on the inflow or outflow in the same time.

Patient follow-up :

Patient follow-up is performed at 1, 6, 12 and 24 months. Follow-up will systematically include a clinical evaluation and a duplex scan with the ankle brachial index (ABI).

The x-rays and the quality of life questionnaire will be done at 1, 12 and 24 months.

All clinical surveillance events, complications and re-hospitalizations will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic PAD, Rutherford 2 to 6
* Atherosclerotic femoropopliteal lesion TASC C or D (on CT scan or arteriography)
* De novo femoropopliteal lesion
* Patient informed of the study and oral authorization collected

Exclusion Criteria:

* Under-age patient
* Patient of age, but under legal guardianship or care
* Potentially pregnant women
* Patients do not understand the French language
* Asymptomatic lesion
* Acute ischemia or acute thrombosis
* Lesion already treated
* No-atherosclerotic disease
* hemostasis disorder
* severe comorbidity with life expectancy less than 2 years
* contraindication of antiplatelet (dual antiplatelet therapy required during at least 2 month post-intervention)
* patient participating in a clinical trial likely to interfer
* Comorbidity or other, according investigator, that may interfere with the conduct of the study
* lesion near to an aneurysm
* Patient follow-up impossible
* Patient refuse to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-05-13 (Estimated); Study Completion 2022-05-13 (Estimated)

PRIMARY OUTCOMES:
Changes in chronic lower limb ischemia at 12 months follow-up | 12 months
  Number of cases of improvement of at least 1 category of Rutherford classification for claudicants.
  Healing of a trophic disorder and disappearance of resting pain for patient with critical ischemia

SECONDARY OUTCOMES:
Changes in chronic lower limb ischemia at 24 months follow-up | 24 months
  Number of cases of improvement of at least 1 category of Rutherford classification for claudicants.
  Healing of a trophic disorder and disappearance of resting pain for patient with critical ischemia
Major adverse cardiovascular events | 24 months
  Number of cases of MACE at 24 months follow-up
Major adverse limb events | 24 months
  Number of cases of MALE at 24 months follow-up
Limb salvage rate | 24 months
  Number of cases of limb salvage at 24 months follow-up
Changes in ankle-brachial index | 24 months
  Changes in mean of ankle-brachial index after procedure at 24 months follow-up
Primary patency | 24 months
  Primary patency rate at 24 months follow-up
Secondary patency | 24 months
  Secondary patency rate at 24 months follow-up
Restenosis rate | 24 months
  Number of cases of significant restenosis (more, than 50%) in stenting arterial segment
Thrombosis rate | 24 months
  Number of cases of thrombosis in stenting arterial segment
Changes in the patients quality of life | 1, 12, 24 months
  Changes in mean of EQ5D-3L questionnaire units after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Alexander A Gostev, Novosibirsk, Novosibirskaya Obl, Russia